CLINICAL TRIAL: NCT00238290
Title: Trastuzumab Monotherapy Followed By the Combination of Trastuzumab and Letrozole in Post-Menopausal Women With ER-Positive, HER-2 Positive Advanced Breast Cancer Resistant to a Nonsteroidal Aromatase Inhibitor: A Multicenter Two-Step Phase II Trial
Brief Title: Trastuzumab and Letrozole in Treating Postmenopausal Women With Progressive Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 23/03; EU-20527
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Experimental): Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes once in weeks 1-3 OR once in week 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression after 9 weeks receive trastuzumab as before and oral letrozole once daily in the absence of further disease progression or unacceptable toxicity.
  Interventions: Drug: Trastuzumab + Letrozole

INTERVENTIONS:
Drug: Trastuzumab + Letrozole — Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes once in weeks 1-3 OR once in week 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression after 9 weeks receive trastuzumab as before and oral letrozole once daily in the absence of further disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. Giving trastuzumab together with letrozole after disease progression may be an effective treatment for breast cancer.

PURPOSE: This phase II trial is studying how well giving trastuzumab together with letrozole works in treating postmenopausal women with progressive advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of trastuzumab (Herceptin®) monotherapy followed by trastuzumab and letrozole in women with progressive advanced breast cancer that is resistant to prior treatment with a nonsteroidal aromatase inhibitor.

Secondary

* Determine the safety profile of this regimen in these patients.
* Correlate HER-2-extracellular domain (ECD) levels with response to treatment in these patients.
* Determine the efficacy of this regimen in these patients.
* Correlate response and time to tumor progression with changes in serum HER-2-ECD levels in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes once in weeks 1-3 OR once in week 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression after 9 weeks receive trastuzumab as before and oral letrozole once daily in the absence of further disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 12 weeks until disease progression and then at 6 months.

PROJECTED ACCRUAL: A total of 30-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Advanced disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion outside previously irradiated areas that is ≥ 20 mm OR ≥ 10 mm if the slice thickness of the CT scan or MRI is ≤ 5 mm

  * No nonmeasurable lesions as the only site of measurable disease, including any of the following:

    * Osteoblastic bone metastases
    * Ascites
    * Pleural or pericardial effusions
    * Carcinomatous lymphangitis of the lung
* Progressive disease after prior treatment with a nonsteroidal aromatase inhibitor (e.g., letrozole or anastrozole) in an adjuvant or advanced disease setting
* HER-2 amplification ≥ 2 by fluorescence in situ hybridization
* No clinical symptoms or history of CNS or leptomeningeal metastases (no imaging is required)
* No visceral involvement with risk for organ dysfunction
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Postmenopausal, defined by 1 of the following:

  * At least 55 years of age
  * Less than 55 years of age with spontaneous cessation of menses for ≥ 1 year
  * Less than 55 years of age with spontaneous cessation of menses within the past year, but amenorrheic with biochemical evidence of postmenopausal status
  * Underwent prior bilateral oophorectomy
  * Radiation or chemically induced menopause (treatment with luteinizing hormone-releasing hormone antagonists must continue during study treatment)

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST and ALT ≤ 2 times upper limit of normal

Renal

* Creatinine clearance > 30 mL/min

Cardiovascular

* No uncontrolled cardiac disease, including any of the following:

  * Unstable angina
  * Arrhythmia
  * Hypertension
* No history of congestive heart failure
* No myocardial infarction within the past 6 months
* LVEF > 50% by echocardiogram

Pulmonary

* No severe dyspnea at rest

Other

* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer
* No psychiatric disability that would preclude study participation or giving informed consent
* No active autoimmune disease
* No uncontrolled diabetes
* No other serious underlying medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior trastuzumab (Herceptin®)

Chemotherapy

* Prior neoadjuvant or adjuvant chemotherapy allowed
* No prior palliative chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* More than 1 month since prior experimental drugs on another clinical trial
* No concurrent drugs that contraindicate study treatment
* No other concurrent anticancer drugs
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-05; Primary Completion 2010-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate as assessed by CT scan or MRI every 3 months | 3 months

SECONDARY OUTCOMES:
Time to tumor progression (TTP) every 3 months | 3 months
Overall survival every 3 months | 3 months
Toxicity every 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koeberle, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (14):
- Switzerland (14):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Ospedale Beata Vergine, Mendrisio
  - Praxis Dr. Beretta, Rheinfelden
  - Kantonsspital - St. Gallen, Sankt Gallen
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Koeberle D, Ruhstaller T, Jost L, Pagani O, Zaman K, von Moos R, Oehlschlegel C, Crowe S, Pilop C, Thuerlimann B; Swiss Group for Clinical Cancer Research (SAKK). Combination of trastuzumab and letrozole after resistance to sequential trastuzumab and aromatase inhibitor monotherapies in patients with estrogen receptor-positive, HER-2-positive advanced breast cancer: a proof-of-concept trial (SAKK 23/03). Endocr Relat Cancer. 2011 Mar 9;18(2):257-64. doi: 10.1530/ERC-10-0317. Print 2011 Apr. PMID 21317203